CLINICAL TRIAL: NCT00050024
Title: The Effect of Peripheral Heterotopic Stimulation on Cortical Excitability in Dystonia
Brief Title: Transcranial Magnetic Stimulation and Electrical Stimulation of Nerves to Study Focal Dystonia
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030048; 03-N-0048
Record Dates: First submitted 2002-11-19; First posted 2002-11-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-09-17

CONDITIONS: Dystonic Disorders
Keywords: TMS; Afferent Stimulation; Motor Cortex; Writer's Cramp; Surround Inhibition; Heterotopic Inhibition; Focal Dystonia; Writer Cramp
MeSH Terms: conditions — Dystonic Disorders

SUMMARY:
This study will use transcranial magnetic stimulation (TMS) and electrical stimulation of nerves to examine how the brain controls muscle movement in focal hand dystonia (writer's cramp). Normally, when a person moves a finger, the brain's motor cortex prevents the other fingers from moving involuntarily. Patients with focal hand dystonia have difficulty with individualized finger movements, possibly due to increased excitability of the motor cortex. Musicians, writers, typists, athletes and others whose work involves frequent repetitive movements may develop focal dystonia of the hand.

Healthy normal volunteers and patients with focal dystonia 18 years of age and older may be eligible for this study.

For the TMS procedure, subjects are seated in a comfortable chair with their hands placed on a pillow on their lap. An insulated wire coil is placed on the scalp. A brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. This may cause muscle, hand or arm twitching if the coil is near the part of the brain that controls movement, or it may induce twitches or transient tingling in the forearm, head or face muscles. Subjects will be asked to move a finger. Just before this movement, a brief electrical stimulation will be applied to the end of either the second or fifth finger. Metal electrodes will be taped to the skin over the muscle for computer recording of the electrical activity of the hand and arm muscles activated by the stimulation. The testing will last 2-3 hours.

...

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effect of sensory afferent input on surround inhibition in the motor cortex in dystonia. Surround inhibition is a cortical phenomenon, the function of which may be to suppress unwanted movements in surrounding muscles during voluntary actions. In support of this, a recent study showed that motor output to the little finger was reduced during self-paced, voluntary movements of the index finger, despite an increase in spinal excitability. Work has also shown that in relaxed muscles, homotopic and heterotopic peripheral stimulation results in time dependent modulation of motor cortical excitability. However, no studies have examined the relationship between volitional movement and sensory input on cortical surround inhibition, the phenomenon which we hypothesize to be defective in dystonia. The aim of this study then is to examine the changes in surround inhibition when electrical stimulation is applied to the finger being actively moved, leading to an inhibition of a surrounding finger (heterotopic inhibition), at different time intervals prior to the initiation of movement, to assess the effect of heterotopic peripheral stimulation on surround inhibition in dystonia patients compared to normal subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:

Nineteen patients age 18 and over with focal dystonia of the upper limbs (writer's cramp) will be recruited for the study.

For patients, the only selection criteria are the presence of focal hand dystonia.

Nineteen normal subjects age 18 and over will be recruited for the control group.

The controls will not have dystonia or any other neurological condition.

All subjects will sign an informed consent prior to participation in the trial.

EXCLUSION CRITERIA:

Exclusion criteria for the trial covering both the normal control and dystonia group will include any concurrent medical or surgical condition as well as neurological or psychiatric illnesses.

Exclusion criteria will include any individual who is on medications with potential influence of the nervous system function (antidepressants, anxiolytics, anticonvulsants, antipsychotic, antiparkinson, hypnotics, stimulants, and antihistamines).

The exclusion criteria also include patients who have received Botulinum toxin injection within 3 months of starting the protocol.

Furthermore, any individual who has a pacemaker, an implanted medical pump, a metal plate or metal object in the skull or eye (for example, after brain surgery), or who has a history of seizure disorder will be excluded from the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38
Dates: Start 2002-11-13; Study Completion 2008-09-17

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Abbruzzese G, Marchese R, Buccolieri A, Gasparetto B, Trompetto C. Abnormalities of sensorimotor integration in focal dystonia: a transcranial magnetic stimulation study. Brain. 2001 Mar;124(Pt 3):537-45. doi: 10.1093/brain/124.3.537. PMID 11222454
- [Background] Hallett M. Transcranial magnetic stimulation and the human brain. Nature. 2000 Jul 13;406(6792):147-50. doi: 10.1038/35018000. PMID 10910346
- [Background] Ahmad F, McPhie P. The denaturation of covalently inhibited swine pepsin. Int J Pept Protein Res. 1978 Sep;12(3):155-63. doi: 10.1111/j.1399-3011.1978.tb02879.x. PMID 29843
- [Background] Hallett M. Is dystonia a sensory disorder? Ann Neurol. 1995 Aug;38(2):139-40. doi: 10.1002/ana.410380203. No abstract available. PMID 7654059